CLINICAL TRIAL: NCT01644136
Title: A Pilot Clinical Trial for the Prevention of Postoperative Lymphoceles Using Absorbable Micorporous Polysaccharide Hemosphere Particles During Robotic Assisted Prostatectomy With Lymph Node Dissection
Brief Title: Microspheres in Preventing Lymphatic Fluid Collection After Surgery in Patients With Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-11017; NCI-2012-00918 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Lymphocele; Prostate Cancer
MeSH Terms: conditions — Lymphocele; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (microsphere-mediated lymphocele prevention) (Experimental): Patients undergo standard robotic assisted laparoscopic prostatectomy with pelvic lymph node dissection. After lymph node dissection, patients undergo microsphere-mediated lymphocele prevention to the lymph node basin on one side of the pelvis.
  Interventions: Procedure: robot-assisted laparoscopic surgery; Procedure: regional lymph node dissection; Device: microsphere-mediated lymphocele prevention

INTERVENTIONS:
Procedure: robot-assisted laparoscopic surgery — Undergo standard robotic assisted laparoscopic prostatectomy
Procedure: regional lymph node dissection — Undergo pelvic lymph node dissection
Device: microsphere-mediated lymphocele prevention — Undergo microsphere-mediated lymphocele prevention

SUMMARY:
This study is being performed to investigate if the application of Arista absorbable hemostat (AH)®, a product approved to stop surgical bleeding, can prevent lymphoceles. Lymphoceles are collections of lymphatic fluid which can occur after a lymph node dissection for cancer. These fluid collections can become symptomatic in some patients. Arista would be applied to one side of the pelvis after a pelvic lymph node dissection, to see if this decreases the number of postoperative lymph fluid collections seen on a computed tomography (CT) scan after surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether, if applied to the lymph node basins after pelvic lymph node dissection, Arista could potentially reduce the formation of lymphoceles and consequently the need for secondary interventions.

OUTLINE:

Patients undergo standard robotic assisted laparoscopic prostatectomy with pelvic lymph node dissection. After lymph node dissection, patients undergo microsphere-mediated lymphocele prevention to the lymph node basin on one side of the pelvis.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Patients with prostate cancer who are electing to undergo robotic radical prostatectomy with pelvic lymph node dissection at The Arthur G. James Cancer Hospital and Solove Research Institute, The Ohio State University Medical Center by Dr. Ronney Abaza

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-07-14 (Actual); Primary Completion 2014-05-06 (Actual); Study Completion 2014-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative lymphocele formation | 3 months after surgery
  The rate of lymphoceles on each side of the pelvis will be compared. Summary statistics will be reported (mean, standard deviation, and range for the continuous variables and frequency and percentages for the categorical variables). In addition, we will determine interrelationships among specific variables using regression and correlation analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ronney Abaza, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu